CLINICAL TRIAL: NCT00302679
Title: Comparison of Colonoscopy and Sigmoidoscopy in Terms of Pain, Acceptance and Procedure Time
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461701245
Record Dates: First submitted 2006-03-12; First posted 2006-03-14 (Estimated); Last update posted 2006-03-14 (Estimated); Status verified 2006-02

CONDITIONS: Pain
Keywords: Colonoscopy; Sigmoidoscopy; Colon cancer screening; Pain; Screening
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
According to experience in a self-payed health check-up center,unsedated total colonoscopy is not inferior or may be better than unsedated sigmoidoscopy in terms of pain and patients' acceptance.

Hypothesis: Unsedated total colonoscopy is not inferior to unsedated sigmoidoscopy in terms of pain and patients' acceptance.

DETAILED DESCRIPTION:
According to American Cancer Society guideline, screening total colonoscopy every 10 years or sigmoidoscopy every 5 years is recommended for average risk people above 50 years old. However,study in Taiwanese population demonstrated that 37.8% of colorectal lesions were beyond reach of sigmoidoscope, and in cases with lesions with advanced pathology, 66.7% did not have distal colorectal lesion. However, many people think colonoscopy is more painful and choose sigmoidoscopy for screening. However, according to experience in a self-payed health check-up center,unsedated total colonoscopy is not inferior or may be better than unsedated sigmoidoscopy in terms of pain and patients' acceptance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who undergo self-payed unsedated colonoscopy or sigmoidoscopy for colon cancer screening.

Exclusion Criteria:

* Difficulty in assessing pain during the procedure and acceptance for the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2006-01; Study Completion 2006-06

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chih Liao, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] 1. Smith RA, Cokkinides V, Eyre HJ. American Cancer Society guidelines for the early detection of cancer, 2004. CA Cancer J Clin 2004;54:41-52. 2. Labianca R, Beretta GD, Mosconi S, Milesi L, Pessi MA. Colorectal cancer: screening. Ann Oncol 2005;16 Suppl 2:ii127-32. 3. Wallace MB, Kemp JA, Trnka YM, Donovan JM, Farraye FA. Is colonoscopy indicated for small adenomas found by screening flexible sigmoidoscopy? Ann Intern Med 1998;129:273-8. 4. Eddy DM. Screening for colorectal cancer. Ann Intern Med 1990;113:373-84. 5. Chiu HM, Wang HP, Lee YC, Huang SP, Lai YP, Shun CT, Chen MF, Wu MS, Lin JT. A prospective study of the frequency and the topographical distribution of colon neoplasia in asymptomatic average-risk Chinese adults as determined by colonoscopic screening. Gastrointest Endosc 2005;61:547-53. 6. Imperiale TF, Wagner DR, Lin CY, Larkin GN, Rogge JD, Ransohoff DF. Risk of advanced proximal neoplasms in asymptomatic adults according to the distal colorectal findings. N Engl J Med 2000;343:169-74. 7. Nicholson FB, Korman MG. Acceptance of flexible sigmoidoscopy and colonoscopy for screening and surveillance in colorectal cancer prevention. J Med Screen 2005;12:89-95.